CLINICAL TRIAL: NCT00256620
Title: Improving Outcomes and Quality of Life After CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 9407000398 Formerly 0794-502CR
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Coronary Artery Bypass Graft Surgery Patients
Keywords: Cardiopulmonary bypass; Coronary artery disease; Cardiac morbidity; Neurologic morbidity; Neurocognitive function; Autoregulation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Mean arterial pressure during cardiopulmonary bypass 80 mmHg vs. customized

SUMMARY:
The principal objective to this randomized trial is to compare the efficacy of two strategies of intra-operative hemodynamic management during cardiopulmonary bypass among patients undergoing primary elective coronary artery bypass graft (CABG) surgery in preventing peri-operative cardiac, cognitive and neurologic morbidity and mortality and post-operative deterioration in the patient's quality of life as measured by the seven domains of SF-36 Health Survey (bodily pain, health perceptions, energy, and mental, physical, social and role function).

DETAILED DESCRIPTION:
In one group, mean arterial pressure (MAP) was 65 mmHg. In the other, the MAP target was determined by the patients usual preoperative MAP. Thus, the trial will evaluate whether tailoring the MAP target for the period of cardiopulmonary bypass to within 10 mmHg of the patients usual MAP, but < 90 mmHg (and thus achieving pressures during bypass within the patients usual autoregulatory range) reduces major neurologic and cardiac morbidity and mortality, as well as cognitive complications, thereby improving post-operative quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary elective/urgent coronary artery bypass graft (CABG) surgery.

Exclusion Criteria:

* Patients who elect not to participate in the study
* Patients undergoing valve replacement or other cardiovascular surgical procedures
* Patients who are not fluent in English
* Patient who cannot provide informed written consent

Ages: 35 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412
Dates: Start 1996-12; Study Completion 1999-12

PRIMARY OUTCOMES:
Quality of life
Cardiac morbidity
Neurologic morbidity
Mortality
Neurocognitive deterioration

SECONDARY OUTCOMES:
• To evaluate the prognostic importance of severe atheromatous disease of the descending aorta as found on transesophageal echocardiography (TEE) as a predictor of neurologic events.
• To correlate TEE and epiaortic scanning for aortic atheroma with transthoracic echocardiography (TTE) in order to develop a non-invasive screening tool.
• To assess the clinical significance of persistent post-operative depression as measured by the CES-D by using a structured clinical interview and to evaluate the relationship between pre-operative depression and the occurrence of cardiac, neurologic a
• To provide data on the mechanism of perioperative neurologic and cognitive complications in order to design other specific intervention to reduce postoperative morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University; Karl Krieger, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States